CLINICAL TRIAL: NCT05625100
Title: Place of Intrathecal CXCL-13 in the Diagnosis of Lyme Neuroborreliosis
Acronym: CXCL13-LYME
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7885
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2022-11

CONDITIONS: Lyme Borreliosis
Keywords: Lyme borreliosis; Lyme neuroborreliosis; Bannwarth syndrome; Intrathecal CXCL-13
MeSH Terms: conditions — Lyme Disease; Lyme Neuroborreliosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuroborreliosis (NBL) is diagnosed in 10-15% of patients with Lyme borreliosis. In Europe in adults, the main clinical manifestation is called "Bannwarth syndrome". This includes painful meningoradiculitis, sometimes accompanied by cranial nerve neuritis. Current European guidelines issued by the European Federation of Neurological Societies (EFNS) recommend the following triad for the diagnosis of "definite NBL": (i) Neurological symptoms suggestive of NBL without any other obvious cause; (ii) CSF pleocytosis; (iii) Intrathecal production of specific anti-Borreliella antibodies. CXCL13, C-X-C chemokine motif ligand 13, is a chemokine implicated in B cell chemotaxis. Extensive literature exists on the analysis of CXCL13i as a diagnostic marker for acute NBL. A recent meta-analysis from 2018, published by Rupprecht et al finds an overall sensitivity and specificity of 89% and 96% respectively, indicating satisfactory diagnostic value. In this study, the investigators wish to assess the place of this new marker in the diagnosis of neuroborreliosis before proposing it as a test carried out by the Borrelia CNR.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject having consulted at the HUS between 01/01/2013 and 31/12/2018
* Subject not having, after being informed, expressed their opposition to the reuse of their data for the purposes of this research

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject under guardianship or curatorship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old) subject having consulted at the HUS between 01/01/2013 and 31/12/2018
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Positivity of the marker (CXCL13-intrathecal) for known cases of NBL and negativity of this one for known non-NBL cases | Files analysed retrospectively from January 01, 2013 to December 31, 2018 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service Laboratoire de Bactériologie - Plateau Technique de Microbiologie - CHU de Strasbourg - France, Strasbourg, France